CLINICAL TRIAL: NCT02715817
Title: The Effect of Virtual Rehabilitation With Nintendo Wii ® and Conventional Therapeutic Exercises in the Treatment of Individuals Post Stroke
Brief Title: Virtual Rehabilitation and Conventional Therapeutic Exercises in the Treatment of Individuals Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Luan Rafael Aguiar dos Santos, Master's Degree student, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 943.738
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Cerebrovascular Disorders
Keywords: Stroke; Hemiparesis; Physical Therapy; Virtual Reality Exposure Therapy; Video Games
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Paresis | interventions — Telerehabilitation; Gait

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual Rehabilitation - VR (Active Comparator): A virtual rehabilitation program (G0) based on the use of the NW for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes.
  The G0 treatment program consists of the following protocols: a) protocol 1 games (Balance Bubble Plus and Tennis); b) protocol 2 games (Rhythm Parade and Boxing).
  Interventions: Other: Virtual Rehabilitation
- Conventional Therapeutic Exercises - CTE (Active Comparator): A program of conventional therapeutic exercises (G1) for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).All treatment groups prior to perform the study interventions,stretches of upper and lower limbs for 10 minutes. The G1 treatment program consists of the following protocols: a) protocol 1: 30 minutes of upper limb PNF diagonal exercise (flexion-abduction-external rotation and extension-abduction-internal rotation), and 10 minutes of scapula PNF diagonal exercise (anterior and posterior elevation); b) protocol 2: 20 minutes of lower limb PNF diagonal exercise (flexion-abduction-external rotation and flexion-abduction-internal rotation),10 minutes of pelvis PNF diagonal exercise (anterior and posterior depression), and 10 minutes gait cycle training;
  Interventions: Other: Conventional therapeutic exercises
- VR and CTE (Experimental): In G2 program will be performed 20 minutes G0 protocol (1 or 2, used alternately between sessions a week) and 20 minutes G1 protocol (1 or 2, used alternately between sessions a week), taking the time of the performed activities halved in both protocols.
  Interventions: Other: Virtual Rehabilitation and Conventional Therapeutic Exercise

INTERVENTIONS:
Other: Virtual Rehabilitation — It is the use of the NW games for rehabilitation of balance and gaite in post-stroke patients.
  Other Names: NW; Non-immersive virtual reality; Commercial Game; Wii-rehabilitation
  Arms: Virtual Rehabilitation - VR
Other: Conventional therapeutic exercises — It is the use of the conventional therapeutic exercises for rehabilitation of balance and gait in post-stroke patients.
  Other Names: Conventional physical therapy; Conventional exercises to improve balance and gait; Diagonals of PNF; PNF method
  Arms: Conventional Therapeutic Exercises - CTE
Other: Virtual Rehabilitation and Conventional Therapeutic Exercise — It is the use of the conventional exercises and of the NW for rehabilitation of balance and gait in post-stroke patients.
  Other Names: Non-immersive virtual reality; Wii-rehabilitation; Commercial Game; Conventional exercises to improve balance and gait; Diagonals of PNF
  Arms: VR and CTE

SUMMARY:
The purpose of this study is to determine the effects of the use the Nintendo Wii® (NW) and conventional therapeutic exercises in the rehabilitation of balance and gait of the post-stroke patients and the impact on quality of life.

DETAILED DESCRIPTION:
This Randomised clinical trial (RCT) has longitudinal and prospective feature, held at the Neurosciences Clinic located at the Clinic Professor Francisco Magalhães Neto the HUPES Complex / Federal University of Bahia from June 2015 until June 2017.

In the initial evaluation were obtained by a trained examiner and blinded to the allocation of participants, all personal data of all patients, as well as evaluations of balance, gait, and quality of life through specific validated scales:

1. Berg Balance Scale (BBS);
2. Tinetti Gait Scale (TGS)
3. Quality of Life Scale Specific for stroke (QLSSS) ;

The investigators employ a program of conventional therapeutic exercises and virtual rehabilitation with NW, for a period of two months, with sessions two times a week for 50 minutes (a total of 16 sessions).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years, of both sexes; clinical diagnosis of stroke confirmed by neurological assessment report or neuroimaging;
* a stroke at least 6 months prior to the study
* the ability to walk independently with or without an assistive device;
* absence of visual or auditory deficits as reported by the subject.

Exclusion Criteria:

* score <24 on the Mini Mental State Examination;
* other associated neurological conditions;
* other orthopedic injuries that could impair mobility and make the execution of the proposed activity impossible;
* participation in other physical rehabilitation programs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
BBS | 8 weeks
  It is a scale that allows a functional assessment of the balance of the performance. It is based on 14 common items of everyday life, graduated from 0 to 4 points, reaching 56 points maximum score.

SECONDARY OUTCOMES:
TGS | 8 weeks
  It is a 12-point instrument of observational analysis of gait ability. The count for each exercise ranges from 0 to 1 or from 0 to 2, with a lower score indicating a poorer physical ability.
QLSSS | 8 weeks
  The QLSS was developed to measure the quality of life of patients with stroke sequela.It contains 49 items arranged into 12 fields, and the score for each item ranges from 1 to 5 points and the total score can range from 49 to 245, so that the lower the score, the greater the degree of dependence and difficult to perform tasks, which indicates a worse perception of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ailton S Melo, PhD, Study Director — Federal University of Bahia
Locations (1):
- Complex Hospital Professor Edgard Santos, Federal University of Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] da Silva Ribeiro NM, Ferraz DD, Pedreira E, Pinheiro I, da Silva Pinto AC, Neto MG, Dos Santos LR, Pozzato MG, Pinho RS, Masruha MR. Virtual rehabilitation via Nintendo Wii(R) and conventional physical therapy effectively treat post-stroke hemiparetic patients. Top Stroke Rehabil. 2015 Aug;22(4):299-305. doi: 10.1179/1074935714Z.0000000017. Epub 2015 Feb 25. PMID 26258455
- [Background] Saposnik G, Teasell R, Mamdani M, Hall J, McIlroy W, Cheung D, Thorpe KE, Cohen LG, Bayley M; Stroke Outcome Research Canada (SORCan) Working Group. Effectiveness of virtual reality using Wii gaming technology in stroke rehabilitation: a pilot randomized clinical trial and proof of principle. Stroke. 2010 Jul;41(7):1477-84. doi: 10.1161/STROKEAHA.110.584979. Epub 2010 May 27. PMID 20508185
- [Background] Saposnik G, Mamdani M, Bayley M, Thorpe KE, Hall J, Cohen LG, Teasell R; EVREST Steering Committee; EVREST Study Group for the Stroke Outcome Research Canada Working Group. Effectiveness of Virtual Reality Exercises in STroke Rehabilitation (EVREST): rationale, design, and protocol of a pilot randomized clinical trial assessing the Wii gaming system. Int J Stroke. 2010 Feb;5(1):47-51. doi: 10.1111/j.1747-4949.2009.00404.x. PMID 20088994
- [Background] Dos Santos LR, Carregosa AA, Masruha MR, Dos Santos PA, Da Silveira Coelho ML, Ferraz DD, Da Silva Ribeiro NM. The Use of Nintendo Wii in the Rehabilitation of Poststroke Patients: A Systematic Review. J Stroke Cerebrovasc Dis. 2015 Oct;24(10):2298-305. doi: 10.1016/j.jstrokecerebrovasdis.2015.06.010. Epub 2015 Aug 21. PMID 26303792
- [Background] Kim K, Lee DK, Jung SI. Effect of coordination movement using the PNF pattern underwater on the balance and gait of stroke patients. J Phys Ther Sci. 2015 Dec;27(12):3699-701. doi: 10.1589/jpts.27.3699. Epub 2015 Dec 28. PMID 26834335
- [Background] Seo K, Park SH, Park K. The effects of stair gait training using proprioceptive neuromuscular facilitation on stroke patients' dynamic balance ability. J Phys Ther Sci. 2015 May;27(5):1459-62. doi: 10.1589/jpts.27.1459. Epub 2015 May 26. PMID 26157240
- See also: World Health Organization. Health topics: Stroke, Cerebrovascular accident. — http://www.who.int/topics/cerebrovascular_accident/en/
- See also: Evidence-Based Review of Stroke Rehabilitation (EBRSR) — http://www.ebrsr.com/